CLINICAL TRIAL: NCT02689154
Title: W8Loss2Go: Behavioral Weight Loss Intervention Utilizing Mobile Health Technology in Pediatric Patients Referred to a Tertiary Care Center Weight Management Clinic
Brief Title: W8Loss2Go: mHealth Weight Management Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Alaina Vidmar, MD, Pediatric Endocrinology Fellow Children's Hospital of Los Angeles, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-16-00007
Record Dates: First submitted 2016-02-15; First posted 2016-02-23 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Pediatric Obesity; Food Addiction; Mobile Health (mHealth); Weight Management
MeSH Terms: conditions — Obesity; Pediatric Obesity; Food Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- W8Loss2Go App (Experimental): Subjects will complete all stages of W8Loss2Go mHealth intervention.
  Interventions: Device: W8Loss2Go

INTERVENTIONS:
Device: W8Loss2Go — The participants will proceed through all parts of the app program (problem food withdrawal, snacking control and withdrawal from excessive portions) and receive weekly phone calls from the study coordinator, who will be monitoring app usage and providing motivation. Subjects will return to the EMPOWER clinic for a three month weight check and face-to-face meeting with their mentor. After the study period, participants will again complete the EBQ, and be offered continued enrollment in the EMPOWER clinic or continued home use of the mHealth technology.

SUMMARY:
The investigators will test a recent mobile technology based (mHealth) behavioral weight loss intervention (W8Loss2Go), which is designed for children and adolescents, and uses an addiction model to promote withdrawal from problem foods, snacking, and excessive amounts at meals. The investigators will test whether this intervention will reduce body mass index (BMI), help subjects identify and withdraw from "problem foods", eliminate snacking, and reduce the amounts of foods consumed at home meals.

DETAILED DESCRIPTION:
Background and Rationale: About one in five 12-18 year-olds in the U.S. are obese. It has been theorized that overeating in some individuals may have addictive qualities, and that specific foods may have addictive potential for these people. But few weight management interventions have tested therapeutic techniques founded in addiction medicine principles to date. Since mHealth interventions have been successful in the treatment of other addictions, the investigators hypothesize that mHealth technologies which are rooted in behavioral theory could be effective to promote weight loss in some individuals.

Dr. Robert Pretlow, together with E-Health International, created a weight loss intervention via an iPhone application (W8Loss2Go), based on the addiction treatment approach of staged, incremental withdrawal from problem foods, snacking/grazing, and excessive amounts of foods at meals. The W8Loss2Go application helps participants address their dependence on specific problem foods prior to addressing the amount of food consumed. A secondary focus of the application is to increase the amount of health provider-patient interaction outside of clinic based face-to-face-sessions in a cost-effective manner. Initial pilot studies in obese adolescents in a community setting showed success in improving these problem behaviors and improving BMI.

Intervention: The investigators will test a recent mobile technology based (mHealth) behavioral weight loss intervention, W8Loss2Go, which is designed for children and adolescents, and uses an addiction model to promote a staged withdrawal from problem foods, snacking, and excessive amounts at meals.

Hypothesis: The investigators hypothesize that participants who display addictive behaviors will respond well the mHealth intervention and will be able to withdraw from problem foods and eliminate snacking and excessive amounts eaten at meals, and will therefore show significant decrease in BMI z score from first to last visit.

Specific Aim 1: Determine if participants utilizing the app can stop eating certain self-identified problem foods.

Specific Aim 2: Determine if participants utilizing the app can reduce the amounts (portion-size and frequency) of foods that they consume in large quantities.

Study Design: New EMPOWER patients complete the Yale Food Addiction Study for Children (YFAS-c), a validated 25 item instrument designed to identify addictive behaviors related to food. Patients with more than two positive criteria on the YFAS-C will be recruited for participation in the W8Loss2Go study. Enrolled subjects and their parents will complete the Eating Behaviors Questionnaire (EBQ-Merlo 2009), and then receive the app, an iPhone 5S (if needed), a wireless body weight scale, and a wireless food scale. Over the next 6 months, subjects will proceed through all parts of the app program (problem food withdrawal, snacking control and withdrawal from excessive portions) and receive weekly phone calls from the study coordinator, who will be monitoring app usage and providing motivation. During the six months study period, subjects will return to the EMPOWER clinic for a three month weight check and face-to face meeting with their mentor. After the study period, participants will again complete the EBQ, and be offered continued enrollment in the EMPOWER clinic or continued home use of the mHealth technology Study Population: Twenty obese 12-18 year old adolescents will be recruited from new patients referred to the CHLA EMPOWER Clinic.

Control Population: The investigators will utilize historical controls using newly referred patients to the EMPOWER clinic who score negative on the YFAS-c.

Methods of Data Analysis: All outcome variables will be compared before and after the intervention using paired t-tests. Further analysis will compare the results of the W8Loss2Go program to the contemporary anthropomorphic changes in patients undergoing standard care in our EMPOWER program, using two sample t-tests.

Significance: This study will evaluate the feasibility of implementing a mHealth intervention in a large clinic setting and further explore the role of food addiction specific weight loss therapies as an effective and sustainable weight management strategy for children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-18 years
2. Patients referred to EMPOWER
3. Positive screen on the Yale Food Addiction Scale for Children
4. Participant will not be leaving the country during the study duration.

Exclusion Criteria:

1. Obesity comorbidities including impaired glucose tolerance, impaired fasting glucose, diabetes, fatty liver with ALT>40, BP > 99th percentile for age, gender, and height
2. Psychiatric illness including depression and anxiety disorder
3. Known developmental delay

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve D Mittelman, MD, PhD, Study Director — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be de-identified and coded. The sponsor of the study will have access to this data through the application download. The data will not be available to the public.

REFERENCES:
- [Background] Chaplais E, Naughton G, Thivel D, Courteix D, Greene D. Smartphone Interventions for Weight Treatment and Behavioral Change in Pediatric Obesity: A Systematic Review. Telemed J E Health. 2015 Oct;21(10):822-30. doi: 10.1089/tmj.2014.0197. Epub 2015 Aug 20. PMID 26290954
- [Background] Dimitrijevic I, Popovic N, Sabljak V, Skodric-Trifunovic V, Dimitrijevic N. Food addiction-diagnosis and treatment. Psychiatr Danub. 2015 Mar;27(1):101-6. PMID 25751444
- [Background] Lin PH, Intille S, Bennett G, Bosworth HB, Corsino L, Voils C, Grambow S, Lazenka T, Batch BC, Tyson C, Svetkey LP. Adaptive intervention design in mobile health: Intervention design and development in the Cell Phone Intervention for You trial. Clin Trials. 2015 Dec;12(6):634-45. doi: 10.1177/1740774515597222. Epub 2015 Jul 30. PMID 26229119
- [Background] Delisle C, Sandin S, Forsum E, Henriksson H, Trolle-Lagerros Y, Larsson C, Maddison R, Ortega FB, Ruiz JR, Silfvernagel K, Timpka T, Lof M. A web- and mobile phone-based intervention to prevent obesity in 4-year-olds (MINISTOP): a population-based randomized controlled trial. BMC Public Health. 2015 Feb 7;15:95. doi: 10.1186/s12889-015-1444-8. PMID 25886009
- [Background] Gearhardt AN, Corbin WR. The role of food addiction in clinical research. Curr Pharm Des. 2011;17(12):1140-2. doi: 10.2174/138161211795656800. PMID 21492090
- [Background] Jeon E, Park HA. Development of a smartphone application for clinical-guideline-based obesity management. Healthc Inform Res. 2015 Jan;21(1):10-20. doi: 10.4258/hir.2015.21.1.10. Epub 2015 Jan 31. PMID 25705553
- [Background] Pretlow RA, Stock CM, Allison S, Roeger L. Treatment of child/adolescent obesity using the addiction model: a smartphone app pilot study. Child Obes. 2015 Jun;11(3):248-59. doi: 10.1089/chi.2014.0124. Epub 2015 Mar 11. PMID 25760813
- [Derived] Vidmar AP, Pretlow R, Borzutzky C, Wee CP, Fox DS, Fink C, Mittelman SD. An addiction model-based mobile health weight loss intervention in adolescents with obesity. Pediatr Obes. 2019 Feb;14(2):e12464. doi: 10.1111/ijpo.12464. Epub 2018 Aug 16. PMID 30117309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 adolescents self-selected into the app intervention. During the intervention period the app participants did not attend the EMPOWER intervention. The app program did not require parental involvement.
Pre-assignment Details: Newly referred patients were pre-screened for eligibility prior to their first clinic visit. YFAS-c was utilized to screen for traits of food addiction. Inclusion criteria included age 12-18 years and positive YFAS-c. Exclusion criteria were: obesity co-morbidities known psychiatric illness or developmental delay, and the inability to read English.
Period: Overall Study
Arm/Group | W8Loss2Go App
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Of the 50 eligible adolescents approached, 18 elected to participate in the app intervention
Arm/Group | W8Loss2Go App
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 14.44 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
zBMI [Mean (Standard Deviation); unit: z-score] — Measure Description: The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A higher number suggests high degree of obesity at baseline.
  z-score | 2.21 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI) z -Score
Description: The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A negative change value reflects a decrease in BMI or a better outcome and a positive change value reflects an increase in BMI or a worsening in the outcome.
Time Frame: Baseline and 6 months
Population: 18 youth that completed the app intervention
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | W8Loss2Go App
Number analyzed (Participants) | 18
z-score | -0.1 (0.04)

2. Secondary Outcome: Number of Participants With Success in Withdrawing From Problem Foods
Description: The number of participants who were able to withdraw from 5 or more problem foods was evaluated.
Time Frame: 6 months
Population: Withdrawal from Problem Food
Measure: Count of Participants; unit: Participants
Arm/Group | W8Loss2Go App
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Number of Participants Able to Eliminated Day Time Snacking
Description: Success in these areas will be determined by data collected from within the application's database.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | W8Loss2Go App
Number analyzed (Participants) | 18
Participants | 18

4. Secondary Outcome: Number of Participants Able to Reduce Daily Meal Portion Size Utilizing Wireless Food Scale.
Description: Success in these areas will be determined by data collected from within the application's database. Participants will weight meals daily and the app will assist the participant in decrease the quantity of food consumed each day until they achieve age appropriate portion size.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | W8Loss2Go App
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: 6 months
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | W8Loss2Go App
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Although these results are encouraging, there are limitations to interpreting these results as they arise from a small, time limited, pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02689154/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02689154/ICF_001.pdf